CLINICAL TRIAL: NCT07046000
Title: Magnetic Resonance Imaging (MRI) Evaluation of Graft Maturation Following Anterior Cruciate Ligament (ACL) Reconstruction With a Connective Tissue Allograft
Brief Title: MRI Evaluation of Graft Maturation Following ACL Reconstruction
Status: Not yet recruiting | Type: Observational
Sponsor: Skye Biologics Holdings, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: SKY-MRI-ACL-01
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: ACL Tears
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACL Reconstruction with Allograft: Subjects who have undergone ACL reconstruction with allograft
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — MRI to assess graft maturation

SUMMARY:
Post-surgical ACL Graft maturation will be assessed at 4.5, 6, 7.5, 9, 10.5, and 12 months with MRI.

ELIGIBILITY:
Inclusion Criteria:

ACL tear and reconstruction; no other knee ligaments needing reconstruction Primary (first-time) ACL tear in the affected knee ACL injury occurred less than 12 months before ACL reconstruction Have no contraindications or allergies to the treatment administered Have current imaging studies (plain radiographs and MRI exams within the past 12 months) of the knee to rule out other etiologic diagnoses Patient underwent ACL reconstruction with a Bone-Patellar Tendon-Bone (BTB) graft harvested from the same knee (ipsilateral autograft) with the Active Matrix tissue Able and willing to comply with the post-operative study follow-up schedule

Exclusion Criteria:

Prior surgery on the index knee within 12 months of enrollment Steroid injection into the index knee within 6 weeks of enrollment Chronic ACL tear whereas the injury occurred more than 12 months ago Multiligamentous injuries whereas any ligament (MCL, PCL, or PLC) in addition to the ACL needs to be reconstructed Patient underwent ACL reconstruction with a hamstring tendon, Achilles tendon or quadriceps tendon graft (any graft other than a patellar tendon BTB) Contraindication to MRI (eg, implanted devices incompatible with MRI). Chrondral lesion of the knee that requires treatment during ACL reconstruction surgery History of advanced osteoarthritis of the knee or patella-femoral joint; KL grade III or higher History of malignant tumor and osseous metastatic disease, History of chronic pain disorders (i.e., fibromyalgia), Current substance abuse (drug or alcohol), by the investigator's judgment, Females who are pregnant, nursing or breastfeeding, or who intend to become pregnant during participation in the study.

Currently participating in, or have been recently exited from (within 30 days from enrollment in this study), or plan to enroll in another clinical study for a bone allograft or drug that may impact participation or outcomes of this study, Currently involved in any injury litigation or workers compensation claims, Has a condition, disorder or other factor that, in the investigator's opinion, would interfere with study participation.

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subject who received primary ACL surgery at Houston Methodist Sugar Land.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Graft Maturation via MRI | From 4.5 months post surgery until 12 months or graft maturation.
  The signal to noise ratio will be calculated at the proximal, mid-substance, and distal positions of the graft

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Sugar Land, Sugar Land, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided